CLINICAL TRIAL: NCT03462589
Title: Randomized, Double-blind, Placebo-controlled, Dose Escalated Tolerance and Pharmacokinetic / Pharmacodynamic Studies of SY-008 Capsules Administered by Chinese Healthy Subjects
Brief Title: Single Ascending Oral Doses of SY-008 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Yabao Pharmaceutical R&D Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SY008001
Record Dates: First submitted 2018-02-11; First posted 2018-03-12 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- SY-008 dose 1 (Experimental): A single dose of SY-008 (2~30mg) taken orally.
  Interventions: Drug: SY-008
- SY-008 dose 2 (Experimental): A single dose of SY-008 (2~30mg) taken orally.
  Interventions: Drug: SY-008
- SY-008 dose 3 (Experimental): A single dose of SY-008 (2~30mg) taken orally.
  Interventions: Drug: SY-008
- SY-008 dose 4 (Experimental): A single dose of SY-008 (2~30mg) taken orally.
  Interventions: Drug: SY-008
- SY-008 dose 5 (Experimental): A single dose of SY-008 (2~30mg) taken orally.
  Interventions: Drug: SY-008
- SY-008 matching placebo (Placebo Comparator): from 6mg to 30mg
  Interventions: Drug: SY-008

INTERVENTIONS:
Drug: SY-008 — The study will be initiated in healthy subjects at a 2-mg dose that is expected to have minimal pharmacologic effect. Doses will be escalated in subsequent dosing process, after appropriate review of safety data. The subsequent planned doses are 6, 12, 18, 24, 30mg successively. The increment of the dose escalation may be reduced, a lower dose may be administered following data review.

SUMMARY:
This is a phase Ⅰ，single-center, randomized, double-blinded, placebo-controlled, single ascending dose trial of SY-008 in healthy subjects.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, dosed tolerability, pharmacokinetic / pharmacodynamic study of a single oral SY-008 capsule for Chinese healthy subjects. Plan to screening total of 54 healthy subjects ， dividing them into 6 dose groups.

ELIGIBILITY:
Inclusion Criteria:

1. Gender: Male and female, gender balance.
2. Age: 18-65 years old (including the boundary values).
3. Weight ≥50kg and 19kg / m2 ≤ BMI ≤ 28kg / m2 [BMI = body weight (kg) / height 2 (m2).
4. fasting plasm glucose (FPG): 3.9-6.1mmol / L (excluding the boundary values).
5. glycosylated hemoglobin (HbA1c) <6.5%.
6. healthy subjects determined by medical history, physical examination, electrocardiogram and laboratory tests. Test results within the normal range for the population or investigator site, or with abnormalities deemed clinically insignificant by the investigator.
7. have venous access sufficient to allow blood sampling as per the protocol.
8. have given written informed consent approved by sponsors and the ethical review board governing the site.
9. are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures.

Exclusion Criteria:

1. are investigator site personnel directly affiliated with this study and their immediate families. Immediate family is defined as a spouse, parent, child or sibling, whether biological or legally adopted.
2. within 3 months prior to screening, complete or withdraw a clinical study, or are currently conducting a clinical study. Or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.
3. have previously completed or withdrawn from this study.
4. 2h postprandial plasm glucose (2hPPG) ≥7.8 mmol / L（Test on -1 Day）.
5. have known allergies to compounds related to SY-008 capsules or multiple drug allergies, or have been treated with SGLT-1(sodium-glucose cotransporter-1) inhibitors in 1 year.
6. have significant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal (such as hemorrhoids, inflammation of GI tract, tumor, history of surgery, habitual bellyache or diarrheal disorders, other motility disorders), endocrine, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs or of constituting a risk when taking the study medication or interfering with the interpretation of data.
7. have a history of alcohol abuse or drug abuse.
8. show evidence or test positive on any of the following: hepatitis B virus surface antigen (HBsAg), hepatitis C virus antibody (HCV), Treponema pallidum antibody (TP), HIV (HIV1 + 2) antibody.
9. have donated blood of 400 mL or more in the last 3 months or provided any blood donation within the last month from screening.
10. are subjects who have an average weekly alcohol intake that exceeds 21 units per week (males) and 14 units per week (females; 1 unit = 12 oz or 360 mL of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits) or are subjects unwilling to stop alcohol consumption 24 hours prior to dosing until the completion of each inpatient study period.
11. consume more than 10 cigarettes per day or the equivalent, or are unable or unwilling to refrain from nicotine during the study.
12. intend to use over-the-counter or prescription medications within 14 days prior to dosing or during the study.
13. subjects not agree to use reliable contraceptive methods (hormones or barriers or abstinence) during the study period and at least 1 month after administration.
14. women were positive for blood pregnancy test within 24 hours prior to enrollment.
15. pregnant or lactating women.
16. in the opinion of the investigator or sponsor, are unsuitable for inclusion in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2018-08-02 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.03 | 7 days
  Number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment.

SECONDARY OUTCOMES:
area under curve (AUC) of SY-008 following oral administration of single ascending dose | 3 days
  to measure the study drug concentration in blood samples to be collected after drug administration.
Cmax of SY-008 following oral administration of single ascending dose | 3 days
  to measure the study drug concentration in blood samples to be collected after drug administration.
T1/2 of SY-008 following oral administration of single ascending dose | 3 days
  to measure the study drug concentration in blood samples to be collected after drug administration.
CL/F (Clearance rectified) of SY-008 following oral administration of single ascending dose | 3 days
  to measure the study drug concentration in blood samples to be collected after drug administration.
glucose levels following single dose of SY-008 | 24 hours
  FPG AUC
insulin secretion following single dose of SY-008 | 3 days
  insulin changes
C-peptide secretion following single dose of SY-008 | 6 hours
  C-peptide change

CONTACTS AND LOCATIONS:
Overall Officials: Feng Shao, Doctor, Principal Investigator — The Frist Affiliated Hospital Of Nanjing Madical University
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No